CLINICAL TRIAL: NCT04764708
Title: Compassion and Metacognition Based Therapy for Schizotypal Personality Disorder: A Pilot Non-inferiority Randomized Controlled Trial on Repeated Measures.
Brief Title: Compassion and Metacognition in Schizotypal Personality
Acronym: CMBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tages Onlus (Other)
Responsible Party: Principal Investigator, Simone Cheli, Principal Investigator, Tages Onlus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 03-07072020
Record Dates: First submitted 2021-02-12; First posted 2021-02-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Schizotypal Personality Disorder
Keywords: schizotypy; psychotherapy; compassion-focused therapy; metacognitively oriented psychotherapy; metacognition; compassion
MeSH Terms: conditions — Schizotypal Personality Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial with Repeated Measures
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Cognitive behavioral therapy plus standard psychopharmacological treatment.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Experimental Group (Experimental): A Third Wave Cognitive Therapy that integrates Compassion Focused Therapy and Metacognitively Oriented Psychotherapy.
  Interventions: Behavioral: Compassion and Metacognition Based Therapy

INTERVENTIONS:
Behavioral: Compassion and Metacognition Based Therapy — The intervention is a Third Wave Cognitive Therapy targeting metacognitive dysfuctions (through Metacognitively Oriented Psychotherapy) and self-criticism (through Compassion Focused Therapy).
  Arms: Experimental Group
Behavioral: Cognitive Behavioral Therapy — Standard Cognitive Behavioral Therapy for Personality Disorders plus Standard Psychopharmacological Treatment.
  Other Names: Standard Psychopharmacological Treatment
  Arms: Control Group

SUMMARY:
The purpose of this study is to assess the safety and efficacy of a newly developed psychotherapy for schizotypal personality disorder. This new form of psychotherapy integrates compassion focused therapy and metacognitively oriented psychotherapy.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a psychological assessment so as to determine eligibility for study entry. Patients who meet the eligibility requirements will be randomized in a double-blind manner in a 1:1 ratio to new integrative psychotherapy or treatment as usual (cognitive behavioral therapy plus standard psychopharmacological treatment). One month after the conclusion of the two forms of treatment (both lasting 6 months), patients will have access to the final follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

- Being diagnosed with Schizotypal Personality Disorder at SCID-5-AMPD

Exclusion Criteria:

* Being under psychotherapy or psychopahrnacological treatment
* Being diagnosed with schizophrenia and other psychotic disorders
* Being diagnosed with bipolar disorder
* Being diagnosed with intelletual disability
* Being diagnosed with any neurological disases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Personality Pathology at 8 months | 9 measurements over the course of 8 months: (i) at 1 month before intervention starts; (ii) once the treatment starts; (iii) 6 measurements at the end of each month of intervention; iv) at 1-month follow-up.
  Decrese of Personality Inventory for DSM-5 - Brief Form (PID-5-BF) total score (with a range of 0 to 75; higher scores indicating a more severe psychopathology) from baseline to final assessment after 8 months.

SECONDARY OUTCOMES:
Schizotypal Personality Disorder Diagnosis (SPD) | Pre-post evaluation between pre-assessment (1-month before the intervention) and 1-month follow-up assessment.
  Recovery from SPD diagnosis at Module III of Structural Clinical Interview for DSM-5 Alternative Model of Personality Disorders (SCID-5-AMPD).
General Psychopathology | Pre-post evaluation between pre-assessment (1-month before the intervention) and 1-month follow-up assessment.
  Decrease of Global Severity Index (with a range of 0 to 4; higher scores indicating a more severe psychopathology) of the Symptom Checklist-90-R (SCL-90-R).
Metacognition | Pre-post evaluation between pre-assessment (1-month before the intervention) and 1-month follow-up assessment.
  Increase of Metacognition Assessment Scale - Abreviated (MAS-A) total score (with a range of 0 to 28; higher scores indicating higher metacognitive functioning).

CONTACTS AND LOCATIONS:
Overall Officials: Simone Cheli, Principal Investigator — Tages Onlus; Gil Goldzweig, Study Chair — The Academic College of Tel-Aviv Yaffo
Locations (1):
- Centro di Psicologia e Psicoterapia Tages Onlus - Firenze, Florence, FI, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual partecipants data underline the results in all the future publications related to the trial will be available after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be released at the end of the study and will be accessible permanently.
Access Criteria: IPD will be accessible on a dedicated web adress inside Tages Onlus website. The page will be released after the end of the study.

REFERENCES:
- [Background] Cheli S, Lysaker PH, Dimaggio G. Metacognitively oriented psychotherapy for schizotypal personality disorder: A two-case series. Personal Ment Health. 2019 Aug;13(3):155-167. doi: 10.1002/pmh.1447. Epub 2019 Jun 6. PMID 31169366
- [Background] Cheli S. Assessment and treatment planning for schizotypal personality disorder: A metacognitively oriented point of view. Psychiatr Rehabil J. 2020 Dec;43(4):335-343. doi: 10.1037/prj0000429. Epub 2020 May 28. PMID 32463252
- [Background] Petrocchi N, Cheli S. The social brain and heart rate variability: Implications for psychotherapy. Psychol Psychother. 2019 Jun;92(2):208-223. doi: 10.1111/papt.12224. Epub 2019 Mar 20. PMID 30891894
- [Background] Lysaker PH, Dimaggio G, Hamm JA, Leonhardt BL, Hochheiser J, Lysaker JT. Disturbances in Self-Experience in Schizophrenia: Metacognition and the Development of an Integrative Recovery-Oriented Individual Psychotherapy. Psychopathology. 2019;52(2):135-142. doi: 10.1159/000495297. Epub 2018 Dec 11. PMID 30537720
- [Background] Dimaggio G, Lysaker PH. Metacognition and mentalizing in the psychotherapy of patients with psychosis and personality disorders. J Clin Psychol. 2015 Feb;71(2):117-24. doi: 10.1002/jclp.22147. Epub 2014 Dec 31. PMID 25557317
- [Background] Lysaker PH, Gagen E, Klion R, Zalzala A, Vohs J, Faith LA, Leonhardt B, Hamm J, Hasson-Ohayon I. Metacognitive Reflection and Insight Therapy: A Recovery-Oriented Treatment Approach for Psychosis. Psychol Res Behav Manag. 2020 Apr 2;13:331-341. doi: 10.2147/PRBM.S198628. eCollection 2020. PMID 32308511
- [Background] Lysaker PH, Hamm JA, Hasson-Ohayon I, Pattison ML, Leonhardt BL. Promoting recovery from severe mental illness: Implications from research on metacognition and metacognitive reflection and insight therapy. World J Psychiatry. 2018 Mar 22;8(1):1-11. doi: 10.5498/wjp.v8.i1.1. eCollection 2018 Mar 22. PMID 29568726
- [Background] Dimaggio G, Semerari A, Carcione A, Procacci M, Nicolo G. Toward a model of self pathology underlying personality disorders: narratives, metacognition, interpersonal cycles and decision-making processes. J Pers Disord. 2006 Dec;20(6):597-617. doi: 10.1521/pedi.2006.20.6.597. PMID 17192140
- [Background] Kramer U, Beuchat H, Grandjean L, Pascual-Leone A. How Personality Disorders Change in Psychotherapy: a Concise Review of Process. Curr Psychiatry Rep. 2020 Jun 9;22(8):41. doi: 10.1007/s11920-020-01162-3. PMID 32519017
- [Background] Heriot-Maitland C, McCarthy-Jones S, Longden E, Gilbert P. Compassion Focused Approaches to Working With Distressing Voices. Front Psychol. 2019 Feb 1;10:152. doi: 10.3389/fpsyg.2019.00152. eCollection 2019. PMID 30774614
- [Background] Kirby JN, Tellegen CL, Steindl SR. A Meta-Analysis of Compassion-Based Interventions: Current State of Knowledge and Future Directions. Behav Ther. 2017 Nov;48(6):778-792. doi: 10.1016/j.beth.2017.06.003. Epub 2017 Jun 21. PMID 29029675
- [Background] Leaviss J, Uttley L. Psychotherapeutic benefits of compassion-focused therapy: an early systematic review. Psychol Med. 2015 Apr;45(5):927-45. doi: 10.1017/S0033291714002141. Epub 2014 Sep 12. PMID 25215860
- [Background] Lucre K, Clapton N. The Compassionate Kitbag: A creative and integrative approach to compassion-focused therapy. Psychol Psychother. 2021 Apr;94 Suppl 2:497-516. doi: 10.1111/papt.12291. Epub 2020 Jul 8. PMID 32639097
- [Background] Braehler C, Gumley A, Harper J, Wallace S, Norrie J, Gilbert P. Exploring change processes in compassion focused therapy in psychosis: results of a feasibility randomized controlled trial. Br J Clin Psychol. 2013 Jun;52(2):199-214. doi: 10.1111/bjc.12009. Epub 2012 Oct 24. PMID 24215148
- [Background] Cohen AS, Mohr C, Ettinger U, Chan RC, Park S. Schizotypy as an organizing framework for social and affective sciences. Schizophr Bull. 2015 Mar;41 Suppl 2(Suppl 2):S427-35. doi: 10.1093/schbul/sbu195. PMID 25810057
- [Background] Debbane M, Eliez S, Badoud D, Conus P, Fluckiger R, Schultze-Lutter F. Developing psychosis and its risk states through the lens of schizotypy. Schizophr Bull. 2015 Mar;41 Suppl 2(Suppl 2):S396-407. doi: 10.1093/schbul/sbu176. Epub 2014 Dec 29. PMID 25548386
- [Background] Mason OJ. The assessment of schizotypy and its clinical relevance. Schizophr Bull. 2015 Mar;41 Suppl 2(Suppl 2):S374-85. doi: 10.1093/schbul/sbu194. PMID 25810054
- [Background] Bora E. Theory of mind and schizotypy: A meta-analysis. Schizophr Res. 2020 Aug;222:97-103. doi: 10.1016/j.schres.2020.04.024. Epub 2020 May 25. PMID 32461089
- [Background] Grant P, Green MJ, Mason OJ. Models of Schizotypy: The Importance of Conceptual Clarity. Schizophr Bull. 2018 Oct 15;44(suppl_2):S556-S563. doi: 10.1093/schbul/sby012. PMID 29474661
- [Background] Kirchner SK, Roeh A, Nolden J, Hasan A. Diagnosis and treatment of schizotypal personality disorder: evidence from a systematic review. NPJ Schizophr. 2018 Oct 3;4(1):20. doi: 10.1038/s41537-018-0062-8. PMID 30282970
- [Background] Rosell DR, Futterman SE, McMaster A, Siever LJ. Schizotypal personality disorder: a current review. Curr Psychiatry Rep. 2014 Jul;16(7):452. doi: 10.1007/s11920-014-0452-1. PMID 24828284
- [Background] Balaratnasingam S, Janca A. Normal personality, personality disorder and psychosis: current views and future perspectives. Curr Opin Psychiatry. 2015 Jan;28(1):30-4. doi: 10.1097/YCO.0000000000000124. PMID 25415496
- [Background] Volkert J, Gablonski TC, Rabung S. Prevalence of personality disorders in the general adult population in Western countries: systematic review and meta-analysis. Br J Psychiatry. 2018 Dec;213(6):709-715. doi: 10.1192/bjp.2018.202. Epub 2018 Sep 28. PMID 30261937
- [Background] Wilson S, Stroud CB, Durbin CE. Interpersonal dysfunction in personality disorders: A meta-analytic review. Psychol Bull. 2017 Jul;143(7):677-734. doi: 10.1037/bul0000101. Epub 2017 Apr 27. PMID 28447827
- [Background] Cheli S, Cavalletti V, Petrocchi N (2020) An online compassion-focused crisis intervention during COVID-19 lockdown: a cases series on patients at high risk for psychosis, Psychosis, 12:4, 359-362, DOI: 10.1080/17522439.2020.1786148
- [Derived] Cheli S, Cavalletti V, Lysaker PH, Dimaggio G, Petrocchi N, Chiarello F, Enzo C, Velicogna F, Mancini F, Goldzweig G. A pilot randomized controlled trial comparing a novel compassion and metacognition approach for schizotypal personality disorder with a combination of cognitive therapy and psychopharmacological treatment. BMC Psychiatry. 2023 Feb 20;23(1):113. doi: 10.1186/s12888-023-04610-5. PMID 36803673

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT04764708/Prot_SAP_ICF_000.pdf